CLINICAL TRIAL: NCT02468128
Title: A Randomized, Double Blind, Placebo-Controlled, Single Dose Study to Assess The Safety and Efficacy of Intramuscular Sebacoyl Dinalbuphine Ester (SDE) for Post-Hemorrhoidectomy Pain Management
Brief Title: A Study of Intramuscular Sebacoyl Dinalbuphine Ester for Post-Hemorrhoidectomy Pain Management
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lumosa Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT1001-301; SDE-2-001 (Other: Taiwan FDA)
Record Dates: First submitted 2015-05-13; First posted 2015-06-10 (Estimated); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Analgesia Disorder; Pain
Keywords: Analgesic; Opioids; Pain relief after surgery; Dinalbuphine; Sebacoyl Dinalbuphine Ester; SDE; SDN; LT1001
MeSH Terms: conditions — Pain | interventions — sebacoyl dinalbuphine ester

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SDE 150mg (Experimental): Single dose, intramuscular, Sebacoyl Dinalbuphine Ester injection 150 mg (2 ml)
  Interventions: Drug: Sebacoyl Dinalbuphine Ester
- placebo (Placebo Comparator): Single dose, intramuscular , Sebacoyl Dinalbuphine Ester placebo injection (2mL)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sebacoyl Dinalbuphine Ester — Intramuscular injection 2mL/vial (75mg/mL)
  Other Names: SDE; LT1001; Nalbuphine Sebacate
  Arms: SDE 150mg
Drug: Placebo — Sebacoyl Dinalbuphine Ester injection placebo, 2mL/vial
  Other Names: Placebo injection
  Arms: placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled, single dose study to assess the safety and efficacy of intramuscular sebacoyl dinalbuphine ester (SDE) for post-hemorrhoidectomy pain management.

DETAILED DESCRIPTION:
This study was a multicenter, double-blind, randomized, placebo-controlled, parallel, pretreatment study, sponsored by Lumosa therapeutics Co., Ltd (Taiwan). All subjects received training of visual analog scores (VAS) before surgery using the 10-mm horizontal version. VAS was taken by study subjects themselves before the first dose of PCA ketorolac, and at 1, 2, 3, 4, 8, 12, 16, 24, 28, 32, 36, 40, 44, 48 hours after surgery. After discharge, VAS was taken, also by the study subjects, twice a day, in the morning and evening of Dayday 3 through Dayday 7. Subjects were asked to complete a short form questionnaire, Brief Pain Inventory, on day 1, day 2, and final visit (day 7-10) after surgery. Patient satisfaction of postsurgical analgesia was assessed at the final visit using a 5-grade categorical scale. The primary objective of the study was to evaluate the efficacy and safety of single intramuscular injection of SDE in an extended-release formulation, against placebo control, administrated pre-operatively in subjects scheduled to undergo elective hemorrhoidectomies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 20 years of age at Screening
* Scheduled to electively undergo 2 or 3-column excisional hemorrhoidectomy
* American Society of Anesthesiology Physical Class 1 - 3
* Adequate clinical lab values (values of potential clinical concern are detailed in Appendix) or, if abnormal, deemed not clinically significant per the Investigator.
* Ability and willingness to provide informed consent, adhere to the study visit schedule and complete all study assessments and language specific questionnaires

Exclusion Criteria:

* Body weight less than 40 kg.
* Concurrent fissurectomy.
* Subject is pregnant or breastfeeding. Women of childbearing potential must have a negative urine pregnancy test at Baseline.
* Women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study.
* History of hypersensitivity or allergy to amide-type local anesthetics, opioid, or any ingredient of the medications administered in this study.
* Subject has a resting respiratory rate less than 8 per minute and blood oxygen saturation less than 90 mmHg.
* Use of any NSAIDs, selective COX-2 inhibitors, opioid, acetaminophen, selective serotonin reuptake inhibitors (SSRI), tricyclic antidepressants (TCA), gabapentin, or pregabalin within three days of surgery.
* Chronic use of opioid medications for more than 14 days in the last 3 months, or non-opioid pain medications more than 5 times per week before screening visit.
* Use of any long-acting opioid medication within 3 days of surgery or any opioid medication within 24 hours of surgery.
* Current painful physical condition or concurrent surgery requires analgesic treatment in the postoperative period.
* Contraindication to epinephrine or any of the pain-control agents planned for postoperative use.
* Administration of an investigational drug within the longer of 30 days or 5 elimination half-lives of such investigational drug prior to study drug administration.
* Any psychiatric disorder, psychological, medical, or laboratory condition that may interfere with study assessments or compliance.
* Significant medical conditions or laboratory results that may indicate an increased vulnerability to study drugs and procedures, and thus expose the subject to an unreasonable risk as a result of participating in this clinical trial.
* Any clinically significant event or condition may be uncovered during surgery.
* History of abuse illicit drugs, prescription medicines or alcohol within the past 2 years.
* Known history of anti-HIV antibody positive
* Failure to pass drug and alcohol screen.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeng-Yi Wang, MD, Principal Investigator — Chang Gung Memorial Hospital-Linkuo
Locations (6):
- Taiwan (6):
  - Chang Gung Memorial Hospital at Chiayi, Chiayi City, Chiayi Hsien
  - Chang Gung Memorial Hospital at Linkou, Linkou District, New Taipei City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung City
  - Chang Gung Memorial Hospital at Keelung, Keelung
  - Cheng Ching General Hospital, Taichung
  - Tri-Service General Hospital, Taipei

REFERENCES:
- [Result] Yeh CY, Jao SW, Chen JS, Fan CW, Chen HH, Hsieh PS, Wu CC, Lee CC, Kuo YH, Hsieh MC, Huang WS, Chung YC, Liou TY, Chiu HH, Tseng WK, Lee KC, Wang JY. Sebacoyl Dinalbuphine Ester Extended-release Injection for Long-acting Analgesia: A Multicenter, Randomized, Double-Blind, And Placebo-controlled Study in Hemorrhoidectomy Patients. Clin J Pain. 2017 May;33(5):429-434. doi: 10.1097/AJP.0000000000000417. PMID 27518486

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled hemorrhoid subjects from 6 sites in Taiwan between 29th December 2012 and 14th April 2015.
Pre-assignment Details: A total of 221 subjects (109 subjects in SDE group; 112 subjects in placebo group) were enrolled into the study and randomized to receive either SDE or placebo treatment.There were 12 of the 221 subjects excluded from the original ITT population since they were protocol violation; therefore, 209 subjects comprised the mITT population.
Period: Overall Study
Arm/Group | SDE 150mg | Placebo
Started | 109 | 112
Completed | 103 | 106
Not Completed | 6 | 6
Not completed — Protocol Violation | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SDE 150mg | Placebo | Total
Number analyzed (Participants) | 103 | 106 | 209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 101 | 104 | 205
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (12.1) | 44.5 (11.4) | 43.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 59 | 111
  Male | 51 | 47 | 98
Region of Enrollment [Number; unit: participants]
  Taiwan | 103 | 106 | 209

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment Calculated as the Area Under the Curve of VAS Pain Intensity Scores Through 48 Hours After Surgery
Description: The primary outcome measure of this study is pain assessment (time-specific pain intensity) calculated as the area under the curve (AUC) of VAS pain intensity scores through 48 hours after surgery (AUC0-48). Pain intensity was measured with visual analog scale (VAS) and the assessment began right before the first use of analgesics, and at 1±0.1, 2±0.1, 3±0.1, 4±0.25, 8±0.5, 12±0.5, 16±0.5, 20±0.5, 24±1, 28±1, 32±2, 36±2, 40±2, 44±2, 48±2 hours after the operation.
Time Frame: 1±0.1, 2±0.1, 3±0.1, 4±0.25, 8±0.5, 12±0.5, 16±0.5, 20±0.5, 24±1, 28±1, 32±2, 36±2, 40±2, 44±2, 48±2 h after the surgery
Population: The analysis included all patients in the modified Intent-to-Treat (mITT) population.
Measure: Mean (Standard Deviation); unit: VAS score*hour
Arm/Group | SDE 150mg | Placebo
Number analyzed (Participants) | 103 | 106
VAS score*hour | 209.93 (111.26) | 253.53 (108.49)
Statistical Analysis 1: Comparison: SDE 150mg vs Placebo; Test type: Superiority or Other; p < 0.01, ANOVA; Mean Difference (Final Values) = -42.20, 95% CI 2-sided [-71.68 to -12.71]

2. Secondary Outcome: Consumption of Ketorolac Via Intravenous Patient- Controlled Analgesia (IV PCA)
Description: Consumption of ketorolac via intravenous Patient- Controlled Analgesia (IV PCA) was calculated through 48 hrs after surgery (study day1-2)
Time Frame: Day 1-2
Population: The analysis included all patients in the modified Intent-to-Treat (mITT) population.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | SDE 150mg | Placebo
Number analyzed (Participants) | 103 | 106
mg | 50.06 (45.72) | 82.33 (66.44)
Statistical Analysis 1: Comparison: SDE 150mg vs Placebo; Test type: Superiority or Other; p < 0.01, ANOVA

3. Secondary Outcome: Pain Assessment Measured With VAS During Day 3-7 in the Morning and Evening, as Well as During Special Events Such as Bowel Movements.
Description: Pain intensity was assessed using a Visual Analog Scale (VAS). The scale ranged from 0 (no pain) to 10 (worst pain imaginable), reported as units on a scale. Higher values indicate worse pain.
  Pain intensity were measured with VAS scores in the morning and evening during Day 3-7.
  It should be noted that the VAS scores during Day 3-7 were not adjusted by rescue medications used for pain relief.
Time Frame: Day 3-7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SDE 150mg | Placebo
Number analyzed (Participants) | 103 | 106
units on a scale
  Day3 Morning | 2.75 (2.30) | 2.79 (2.28)
  Day3 Evening | 3.51 (2.80) | 3.39 (2.75)
  Day4 Morning | 3.30 (2.46) | 3.78 (2.73)
  Day4 Evening | 3.27 (2.69) | 3.56 (2.67)
  Day5 Morning | 3.05 (2.54) | 3.46 (2.51)
  Day5 Evening | 3.20 (2.72) | 3.38 (2.60)
  Day6 Morning | 2.88 (2.51) | 3.20 (2.66)
  Day6 Evening | 2.67 (2.36) | 3.08 (2.63)
  Day7 Morning | 2.50 (2.33) | 2.98 (2.60)
Statistical Analysis 1: Comparison: SDE 150mg vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

4. Secondary Outcome: Time From the End of Operation to the First PCA Ketorolac Dose
Time Frame: From the end of operation until the first PCA ketorolac dose used, assessed up to 48 hrs
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | SDE 150mg | Placebo
Number analyzed (Participants) | 103 | 106
hours | 4.67 [3.58 to 6.73] | 4.32 [2.43 to 5.00]
Statistical Analysis 1: Comparison: SDE 150mg; Test type: Superiority or Other; p < 0.05, Log-rank tests; Log-rank tests were used to compare SDE and placebo with respect to the distribution of time to first post-surgical usage of ketorolac medication

5. Secondary Outcome: Brief Pain Inventory (BPI)
Description: Pain severity was assessed using the Brief Pain Inventory (BPI). The BPI pain severity score is based on a numeric rating scale ranging from 0 to 10 units on a scale, where 0 indicates no pain and 10 indicates pain as bad as you can imagine. Higher scores represent worse pain outcomes. Assessments were conducted on Day 1, Day 2, and Day 7.
Time Frame: Day 1, 2 and Day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SDE 150mg | Placebo
Number analyzed (Participants) | 103 | 106
units on a scale
  Day1 | 3.50 (2.54) | 3.60 (2.24)
  Day2 | 3.14 (2.34) | 3.20 (2.07)
  Day7 | 2.94 (2.10) | 3.19 (2.20)
Statistical Analysis 1: Comparison: SDE 150mg vs Placebo; ANOVA with Treatment, Center effect (and Treatment*Center effect if p-value ≤ 0.1 in non-reduced model); Test type: Superiority — ANOVA with Treatment, Center effect (and Treatment*Center effect if p-value ≤ 0.1 in non-reduced model); p < 0.05, ANOVA — ANOVA with Treatment, Center effect (and Treatment*Center effect if p-value ≤ 0.1 in non-reduced model); ANOVA with Treatment, Center effect (and Treatment*Center effect if p-value ≤ 0.1 in non-reduced model)

6. Secondary Outcome: Consumption of Oral Ketorolac (Day 3-7)
Description: Patients discharged on Day 2. The total amount of oral Ketorolac, as supplemental analgesics after discharge, was used to evaluate the efficacy of extended-release SDE compared with the placebo group.
Time Frame: Day 3-7
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | SDE 150mg | Placebo
Number analyzed (Participants) | 103 | 106
mg | 3.86 (0.81) | 4.29 (0.69)
Statistical Analysis 1: Comparison: SDE 150mg vs Placebo; Test type: Superiority or Other; p < 0.01, ANOVA

7. Secondary Outcome: Subject Satisfaction With Post-Surgical Analgesic Between Treatment Groups
Description: Subject will be asked to classify themselves as either: 'highly satisfied', 'satisfied', 'uncertain', 'dissatisfied' or 'very dissatisfied' at final visit, and a Cochran-Mantel-Haenszel test was used in comparison of subjects' satisfaction with post-surgical analgesic between treatment groups.
Time Frame: Day 7
Measure: Number; unit: participants
Arm/Group | SDE 150mg | Placebo
Number analyzed (Participants) | 102 | 106
participants
  Highly satisfied | 18 | 20
  Satisfied | 68 | 69
  Uncertain | 13 | 10
  Dissatisfied | 3 | 6
  Very dissatisfied | 0 | 1
Statistical Analysis 1: Comparison: SDE 150mg vs Placebo; At the final visit, each subject was asked the questions for evaluation of satisfaction and a Cochran-Mantel-Haenszel test was used in comparison of subjects' satisfaction with post-surgical analgesic between treatment groups; Test type: Superiority or Other — At the final visit, each subject was asked the questions for evaluation of satisfaction and a Cochran-Mantel-Haenszel test was used in comparison of subjects' satisfaction with post-surgical analgesic between treatment groups; p > 0.05, Cochran-Mantel-Haenszel — Satisfaction was evaluated using a patient-reported rating scale to assess the subject's overall satisfaction with postoperative analgesia. More participants indicate greater satisfaction with that treatment

8. Post Hoc Outcome: Post-hoc Analysis of Secondary Outcome Measures (Pain Assessment During Day 3-7)
Description: Pain assessment during Day 3-7 was not corrected for the use of rescue medication in the initial secondary endpoint analysis as that was done for the primary end point, where the VAS scores for the measurement of pain intensity from 0 to 48 hours post-surgery were calculated as the area under the curve (AUC0-48). And for the calculation of AUC, data were imputed with the use of the windowed worst observation carried forward plus last observation carried forward method.For subjects who used rescue medication for pain relief, their VAS scores recorded within the window of ketorolac medication (6 hours, which is one half-life of ketorolac) was replaced by the "worst" observation (i.e., the highest score before taking ketorolac). For the post hoc analysis, the same principle was applied, i.e. the VAS scores AUC0-final (Time zero post-surgery to final visit) were analyzed following the same methodology used for AUC0-48
Time Frame: Day 3-7
Measure: Mean (Standard Deviation); unit: VAS score*hour
Arm/Group | SDE 150mg | Placebo
Number analyzed (Participants) | 103 | 106
VAS score*hour | 630.79 (350.90) | 749.94 (353.72)
Statistical Analysis 1: Comparison: SDE 150mg vs Placebo; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Final Values) = -115.20, 95% CI 2-sided [-209.153 to -21.26]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | SDE 150mg | Placebo
Serious Adverse Events (participants affected / at risk) | 8/109 | 2/112
Other Adverse Events (participants affected / at risk) | 76/109 | 62/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SDE 150mg (N=109) | Placebo (N=112)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urine retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 0 (0)
Injection site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SDE 150mg (N=109) | Placebo (N=112)
Pyrexia (General disorders) | 41 | 20
Constipation (Gastrointestinal disorders) | 13 | 12
Dysuria (Renal and urinary disorders) | 12 | 11
Dizziness (Nervous system disorders) | 18 | 4
Vomiting (Gastrointestinal disorders) | 10 | 1
Nausea (Gastrointestinal disorders) | 5 | 3
Urinary retention (Renal and urinary disorders) | 6 | 6
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 7
Injection site reaction (General disorders) | 34 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days